CLINICAL TRIAL: NCT04682210
Title: A Phase III, Randomized, Open-lable, Multi Center Study of Sintilimab Plus Bevacizumab Versus Active Surveillance as Adjuvant Therapy in Patients With Hepatocellular Carcinoma at High Risk of Recurrence After Curative Hepatic Resection
Brief Title: Sintilimab Plus Bevacizumab as Adjuvant Therapy in HCC Patients at High Risk of Recurrence After Curative Resection
Acronym: DaDaLi
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, MD, Department of Hepatobilliary Surgery, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-280-01
Record Dates: First submitted 2020-12-20; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: HCC; Adjuvant Therapy; Immunotherapy
MeSH Terms: interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): sintilimab 200mg + bevacizumab 7.5mg/kg IV Q3W
  Interventions: Drug: Sintilimab; Drug: Bevacizumab
- Arm B (No Intervention): Active surveillance

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg IV Q3W
  Other Names: Tyvyt
  Arms: Arm A
Drug: Bevacizumab — Bevacizumab 7.5mg/kg IV Q3W
  Other Names: Byvasda
  Arms: Arm A

SUMMARY:
This is an open label, multi-center, randomized, controlled phase III study, to evaluate the efficacy and safety of sintilimab plus bevacizumab as adjuvant therapy in hepatocellular carcinoma (HCC) patients who are at high risk of recurrence after radical resection

DETAILED DESCRIPTION:
There is no stardard adjuvant treatment for HCC. This study is to to evaluate the efficacy and safety of sintilimab plus bevacizumab as adjuvant therapy in HCC patients who are at high risk of recurrence after radical resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first diagnosis of HCC who have undergone a curative resection
* Radiologic evidence of disease free ≥4 weeks after complete surgical resection
* Full recovery from surgical resection or post-operative transarterial chemoembolization before randomization
* Randomization needs to occur within 12 weeks of the date of surgical resection
* High risk for HCC recurrence as protocol defined
* Child-Pugh Score, Class A
* ECOG performance status 0 or 1
* No prior systemic anticancer therapy for HCC
* Adequate hematologic and organ function

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC
* Evidence of residual, recurrent, or metastatic disease at randomization
* History of hepatic encephalopathy or organ transplantation
* Patients who are in the waiting list for liver transplantation
* Patients with Vp4 portal vein thrombosis
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or other immunotherapy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival (RFS) | up to 36 months after randomization
  RFS is defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC as determined by the investigator, or death due to any cause (whichever occurs first).

SECONDARY OUTCOMES:
Overall Survival (OS） | up to 48 months after randomization
  OS is defined as the time from the date of randomisation until death due to any cause
RFS Rate at 12 and 24 months | at 12 and 24 months after randomization
  RFS rate defined as the proportion of patients without recurrence or death from any cause at 12 and 24 months after randomization.
OS Rate at 24 and 36 Months | at 24 and 36 months after randomization
  OS rate defined as the proportion of patients who have not experienced death from any cause at 24 and 36 months after randomization.
TTR(time to recurrence) | up to 36 months after randomization
  TTR is defined as the time the date of randomisation until first documented disease recurrence.
Adverse Events (AEs) | up to 48 months after randomization
  The grade of AEs and the number of patients with AEs are assessed by the investigator based on CTCAE v5.0 from the date of randomization to 90 days after last dose of study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided